CLINICAL TRIAL: NCT05056844
Title: Contrast Enhanced Spectral Mammography (CESM) for the Evaluation of Pathologic Nipple Discharge: A Pilot Study
Brief Title: Contrast Enhanced Spectral Mammography for the Evaluation of Pathologic Nipple Discharge
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2021-0025; NCI-2021-07594 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2021-0025 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2021-09-07; First posted 2021-09-27 (Actual); Last update posted 2025-10-09 (Actual); Status verified 2025-10

CONDITIONS: Breast Carcinoma
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Diagnostic (CESM, DBT) (Experimental): Patients receive iodine-based contrast agent IV then undergo CESM over 10-15 minutes. Patients who have not undergone standard of care DBT within 3 months from the study, also undergo DBT.
  Interventions: Procedure: Contrast Enhanced Digital Mammography; Procedure: Digital Tomosynthesis Mammography; Drug: Iodinated Contrast Agent; Other: Questionnaire Administration

INTERVENTIONS:
Procedure: Contrast Enhanced Digital Mammography — Undergo CESM
  Other Names: CEDM; Contrast Enhanced Spectral Mammography; Contrast-Enhanced Digital Mammography; Contrast Enhanced Mammography
Procedure: Digital Tomosynthesis Mammography — Undergo DBT
  Other Names: DBT; Digital Breast Tomosynthesis; Digital Tomosynthesis of the Breast
Drug: Iodinated Contrast Agent — Given iodine-based contrast agent IV
  Other Names: Iodinated Contrast Dye; Iodine-containing Contrast Media
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This clinical trial studies contrast enhanced spectral mammography (CESM) for the evaluation of pathologic nipple discharge. CESM is similar to standard mammography, but it includes an intravenous (by vein) injection of an iodine-based contrast, which makes tissue and blood vessels more visible in scans. The goal of this trial is to learn if CESM, is better than standard mammography in quickly and efficiently determining the cause of nipple discharge and detecting breast cancer, if present. CESM may increase the chance of finding breast cancers and lower the risk of having unnecessary biopsies.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the added sensitivity of contrast enhancement of CESM (represented by the subtracted contrast images of CESM) compared to low energy [LE] images of CESM (full field digital mammogram [FFDM] equivalent) in detecting the causative lesion (invasive malignancy, ductal carcinoma in situ [DCIS], atypia, or papilloma) in patients with pathologic nipple discharge (PND).

SECONDARY OBJECTIVES:

I. To compare the sensitivity, specificity, negative predictive value, and positive predictive value of CESM versus DBT and ultrasound (US) in predicting invasive malignancy or DCIS in patients with PND.

II. To compare the accuracy of digital breast tomosynthesis (DBT) and LE in the detection of invasive malignancy or DCIS, as well as in the detection of the causative lesion.

III. To estimate the proportion of cases in which CESM affects the choice of the lesion targeted for a biopsy with any imaging modality.

IV. To evaluate the cancer detection rate and the outcomes (need for additional imaging, biopsies, and final pathologic results) of incidental CESM findings.

EXPLORATORY OBJECTIVES:

I. To evaluate the correlation of blood biomarkers and the presence of invasive cancer and DCIS on pathology in the study patients.

II. To evaluate the role of the CESM enhancement pattern in choosing a precise target for a stereotactic biopsy.

III. To evaluate the effect of CESM on the patient workflow by calculating the time from presentation to the definitive diagnosis.

IV. To evaluate the technical feasibility of using CESM- guided or CESM directed biopsies.

V. In patients who undergo a CESM targeted or CESM directed biopsy we will evaluate the upgrade rate of DCIS to invasive malignancy or high-risk lesions to in-situ or invasive cancer for those patients who will require surgery as a part of their routine clinical care.

VI. In those study patients who undergo breast MRI as a part of their clinical care, the sensitivity and specificity of magnetic resonance imaging (MRI) and CESM for the detection of causative lesions will be compared.

OUTLINE:

Patients receive iodine-based contrast agent intravenously (IV) then undergo CESM over 10-15 minutes. Patients who have not undergone standard of care DBT within 3 months from the study, also undergo DBT.

ELIGIBILITY:
Inclusion Criteria:

* Women presenting to MDACC for the evaluation of PND as the main or accompanying symptom
* Age 25-85 years
* Willing to participate in the study and undergo an IV placement, able to undergo iodinated contrast injection, and able to provide informed consent

Exclusion Criteria:

* Reported history of an allergic reaction to iodinated contrast
* History of anaphylactic reaction to any substance in the absence of a prior history of uneventful administration of iodine-based IV contrast.
* Renal insufficiency
* Pregnancy or lactation within 6 months
* Breast surgery affecting the symptomatic breast within prior 6 months, if it was located within 5 cm from the nipple
* Breast biopsy of the symptomatic breast within the last 2 months, if it was located within 5 cm from the nipple
* Breast MRI performed within 24 months before the patient presented with qualifying symptoms (MRI performed contemporarily with CEM for the evaluation of new symptoms is not an exclusion criterion).
* Known breast cancer or active inflammatory process (such as abscess or mastitis) in the breast of concern

Ages: 25 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2021-04-15 (Actual); Primary Completion 2027-04-30 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Sensitivity of contrast enhancement of contrast enhanced spectral mammography (CESM) | through study completion, an average of 1 year
  Will be compared to low exposure (LE) images of CESM (full field digital mammogram equivalent) in detecting the causative lesion (invasive malignancy, ductal carcinoma in situ (DCIS), atypia, or papilloma) in patients with pathologic nipple discharge (PND).

CONTACTS AND LOCATIONS:
Overall Officials: Olena Weaver, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org